CLINICAL TRIAL: NCT05731661
Title: Optimize the Support of Patients in Pelvic Onco-gynecology Through Adapted Support Care in the Post-cancer Period. AFTERGYN Pilot Phase
Acronym: AFTERGYN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-A01872-41
Record Dates: First submitted 2023-01-23; First posted 2023-02-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Long Term Cancer Side Effects; Supportive Care in Cancer; Cancer Survivorship Care Plan; Advanced Nurse Practitioner; Pelvic Gynecological Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delivery of a Personalized Post-Cancer Plan (PPAC) with a day hospitalization in supportive care (Experimental)
  Interventions: Other: Day hospitalization in support care with meeting with support care professionals and coordination of actions by the advanced practice nurse; Other: Delivery of a personalized post-cancer plan
- Delivery of a Personalized Post-Cancer Plan (PPAC) without day hospitalization in supportive care (Active Comparator)
  Interventions: Other: Delivery of useful information according to support care needs, concerning support care professionals in the city; Other: Delivery of a personalized post-cancer plan
- Observational cohort (Other)
  Interventions: Other: Delivery of a personalized post-cancer plan

INTERVENTIONS:
Other: Day hospitalization in support care with meeting with support care professionals and coordination of actions by the advanced practice nurse — During this day hospitalization, patients will meet with different specialized professionals depending on the support care needs identified.
  Arms: Delivery of a Personalized Post-Cancer Plan (PPAC) with a day hospitalization in supportive care
Other: Delivery of useful information according to support care needs, concerning support care professionals in the city — Delivery of useful information according to support care needs, concerning support care professionals in the city
  Arms: Delivery of a Personalized Post-Cancer Plan (PPAC) without day hospitalization in supportive care
Other: Delivery of a personalized post-cancer plan — Delivery of a personalized post-cancer plan

SUMMARY:
While the sequelae and toxicities after ovarian and endometrial cancer treatments are well described in the literature, the actual needs of patients for supportive oncology care remain poorly documented. Moreover, there is no data available to estimate the complexity of the oncological support care actions to be implemented.

It is expected that an evaluation of the needs for supportive oncology care and its organization in day hospitalization for supportive oncology care will lead to an improvement in personalized post-cancer follow-up for these patients and to an improvement in their long-term quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient in complete remission after first-line treatment for endometrial or ovarian/fallopian tube/peritoneal cancer
* Patient having completed her initial treatment; patients with maintenance treatments are eligible
* Mastery of the French language
* Patient with a telephone line
* Patient affiliated to a social security scheme
* Signature of informed consent before any specific procedure related to the study

Exclusion Criteria:

* Any associated medical or psychiatric conditions that could compromise the patient's ability to participate in the study
* Patient with locoregional or metastatic recurrence
* Patient deprived of liberty, under guardianship or curatorship
* Simultaneous participation in a therapeutic clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who used at least one of the oncology support services recommended in the Personalized After-Cancer Care Plan within 4 months of receiving the Personalized After-Cancer Care Plan | Up to 4 months

SECONDARY OUTCOMES:
Proportion of patients with sequelae after the initial treatment of their cancer, as well as the type and grade of the sequelae, based on the National Cancer Institute's screening grids (levels 1 and 2) during the consultation with a nurse referent | Up to 4 months
Description of the types of oncological support care needs identified | Up to 4 months
Proportion of patients with identified cancer care needs (at least one cancer care need to be implemented) 4 months after the submission of the Personalized Cancer Care Plan | Up to 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No